CLINICAL TRIAL: NCT02074241
Title: Molecular Markers of Chemosensitivity for Locally Advanced, Recurrent and Metastatic Bladder Cancer Based on the Adjuvant Chemotherapy of Gemcitabine and Cisplatin-a Prospective Control Study
Brief Title: Molecular Markers of Chemosensitivity for Bladder Cancer
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Zhiwen Chen, M.D,Ph.D, Southwest Hospital, China
Other Study IDs: 2012XLC02-2; 2012XLC02 (Other Grant/Funding Number: 2012XLC02,Third Military Medical University，China)
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Bladder Cancer; Effects of Chemotherapy
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bladder cancer specimens
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Positive Expression: Expression analysis:Positive expression of DNA repair-related genes(XPC, XPF, Brca1, Rad51,SNF5, etc) in bladder cancer specimens.
  Interventions: Other: Expression analysis
- Negative Expression: Expression analysis:Negative expression of DNA repair-related genes(XPC, XPF, Brca1, Rad51, SNF5,etc) in bladder cancer specimens.
  Interventions: Other: Expression analysis

INTERVENTIONS:
Other: Expression analysis — Analysis of the expression of DNA repair genes (XPC, XPF, Brca1, Rad51,SNF5, etc.) in bladder cancer specimens.
  Other Names: E-A

SUMMARY:
The purpose of this study is to try to figure out some bio-markers of chemosensitivity for adjuvant chemotherapy for bladder cancer.

DETAILED DESCRIPTION:
Figure out some bio-markers of chemosensitivity for adjuvant chemotherapy for bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years of age or older, estimated life expectancy ≥ 6 months.
2. .Gone through standardize radical cystectomy and pelvic lymphadenectomy or inoperable.
3. Transitional cell carcinoma of bladder, stage pT3N0M0,T2N1M0-T3-4N1-2M1.Transitional cell carcinoma may be with or without squamous cell carcinoma and/or adenocarcinoma components.
4. Electrocorticography(ECOG) performance status 0-2.
5. Blood routine:Absolute neutrophil count (ANC) ≥ 1500/μL,White blood cell count ≥ 3000/μLPlatelets ≥ 100,000/μL,Hemoglobin ≥ 10.0 g/dL,
6. Total serum bilirubin≤ 1.5 x upper limit of normal (ULN).Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase(SGOT)) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase (SGPT)) ≤ 2.5 x upper limit of normal (ULN).
7. Creatinine clearance rate,Ccr ≥ 60%
8. ECG：no arrhythmias, no myocardial infarction. Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment.

Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests,and other study procedures.

Exclusion Criteria:

1. Past history of systemic chemotherapy
2. Serious heart and lung dysfunction.
3. Associated with central or peripheral neuropathy greater than 2 grade.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. The patients of locally advanced, recurrent, metastatic transitional cell carcinoma.
  2. Gone through standardize radical cystectomy and pelvic lymphadenectomy or inoperable.
  3. Experienced adjuvant chemotherapy(Gemcitabine and Cisplatin).
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-03; Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
cancer progressive free survival rate | 60 months

SECONDARY OUTCOMES:
overall survival | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhiwen Chen, M.D,Ph.D, Principal Investigator — Southwest Hospital, China
Locations (1):
- Southwest hospital,Chian, Chongqing, Chongqing Municipality, China